CLINICAL TRIAL: NCT01791192
Title: A Multicenter, Randomized, Active-controlled Study to Assess the Safety, Tolerability, and Efficacy of FTY720 in Patients With Acute, Noninfectious Intermediate, Posterior and Pan Uveitis
Brief Title: Study of FTY720 in Patients With Uveitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFTY720D2205; 2011-004160-30 (EudraCT Number)
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2014-04

CONDITIONS: Acute Noninfectious Posterior, Intermediate, or Pan Uveitis
Keywords: Uveitis, Fingolimod, Phase II, Visual Acuity, Vitreous Haze, OCT
MeSH Terms: conditions — Uveitis; Ornithine Carbamoyltransferase Deficiency Disease | interventions — Fingolimod Hydrochloride; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FTY720 (Experimental): Fingolimod
  Interventions: Drug: FTY720
- Oral Corticosteroid (Active Comparator): Oral Corticosteroid
  Interventions: Drug: Oral Corticosteroid

INTERVENTIONS:
Drug: FTY720 — Fingolimod
  Arms: FTY720
Drug: Oral Corticosteroid — Oral Corticosteroid
  Arms: Oral Corticosteroid

SUMMARY:
This study will assess the safety, tolerability, and efficacy of FTY720 in patients with acute, noninfectious intermediate, posterior and pan uveitis

ELIGIBILITY:
Inclusion Criteria:

* Acute noninfectious posterior, intermediate, or pan uveitis
* Vitreous haze score of 1+ or more in the study eye at screening and baseline visits

Exclusion Criteria:

* Vaso-occlusive vasculitis involving the retinal macula
* Behçet's uveitis
* Patients requiring corticosteroid or another systemic immunosuppressive medication for any other disease (e.g., asthma or some other autoimmune disease) that would contraindicate tapering (topical steroids permitted)
* Other protocol defined inclusions and/or exclusions may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change in Vitreous Haze Score in the Study Eye at Day 8 | Day 8
  On day 8 of the study, the vitreous haze score will be measured in patients during a dilated fundus examination (using eye drops to enlarge the pupil of the eye). The ophthalmologist will examine the back of the eye to obtain this measure.

SECONDARY OUTCOMES:
Change in Vitreous Haze Score in the Study Eye on Study Examination Days | Days 2, 4, 29, 57
  On study examination days, the vitreous haze score will be measured in patients during a dilated fundus examination (using eye drops to enlarge the pupil of the eye). The ophthalmologist will examine the back of the eye to obtain this measure.
Changes in Visual Acuity (Number of letters) in the Right and Left Eyes on Study Examination Days | Days 2, 4, 8, 29 and 57
  Change in visual acuity will be assessed in the right and left eyes using the ETDRS (early treatment diabetic retinopathy study) visual acuity charts. Change in acuity is defined as the change in the number of letters correctly read on each chart.
Changes in Macular Thickness (Thickness at the Center of the Retina) in the Right and Left Eyes on Study Examination Days | Days 2, 4, 8, 29 and 57
  Macular thickness will be measured using an OCT (optical coherence tomography or type of ultrasound of the eye) on the right and left eyes. This test measures how thick the retina is; the study measure is the thickness at the central part of the eye.
Measures of the Safety and Tolerability of the Study Medication FTY720; Also Measures of Whether the Patients Required Rescue Medication for their Uveitis. | Days 2, 4, 8, 29 and 57
  This will be determined by how safe the study medication FTY720 is determined to be, by how well tolerated it is by the patients and also by whether the patients needed rescue medication (e.g. other medication to treat their uveitis if the study drug was not effective during the time they received it).
Levels of FTY720 and FTY720-P Blood Concentrations Measured in the Patients on Study Examination Days | Days 2, 29 and 57
  The blood FTY720 and FTY720-P concentrations will be measured by collection of 3 mL of blood taken from the patients during specified study examination visits.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals